CLINICAL TRIAL: NCT01505699
Title: Micro RNA Expression Analysis in B-Lineage Adult Acute Lymphoblastic Leukemia From ALL Trial, E2993, Including Patients With Various Cytogenetic and Molecular Abnormalities
Brief Title: Biomarkers in Samples From Patients With B-Cell Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000720304; ECOG-E2993T4
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Leukemia
Keywords: adult acute lymphoblastic leukemia in remission; B-cell adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Cytogenetic Analysis; Microarray Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: RNA analysis
Genetic: cytogenetic analysis
Genetic: microarray analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in samples from patients with acute lymphoblastic leukemia enrolled on ECOG-2993 clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify microRNAs that behave as oncogenes or as tumor suppressor genes in B-lineage acute lymphoblastic leukemia (ALL) in vitro and in vivo.
* To examine if single microRNA or signatures of microRNA correspond to different clinical outcomes in cytogenetically distinct B-ALL groups.

OUTLINE: RNA from archived samples are analyzed for microRNA expression profile in vitro and in vivo.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Samples from patients enrolled on ECOG-2993
* Samples from patients with recurrent cytogenetic abnormalities other than BCR-ABL, including MLL/AF4, E2A/PBX1, and TEL/AML1

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Samples from patients enrolled on E2993 who provided samples for research
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2012-01-06 (Actual); Primary Completion 2012-02-06 (Actual); Study Completion 2012-02-06 (Actual)

PRIMARY OUTCOMES:
Comprehensive view of microRNA expression by cytogenetic subgroup | 1 year
MicroRNA expression in relation to clinical outcome | 1 year
Differential microRNA expression between normal B-cells and progenitors compared to B-ALL | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Guido Wendel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center